CLINICAL TRIAL: NCT06859385
Title: Investigation of the Validity and Reliability of the Standing Up From Supine Test in Parkinson's Patients
Brief Title: Validity and Reliability of the Standing Up From Supine Test With Parkinson's Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, Physiotherapy and Rehabilitation Department, Assistant Professor, Sanko University
Other Study IDs: hakanpolat2
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Parkinson
Keywords: parkinson

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In individuals diagnosed with Parkinson's disease, not being able to stand up especially after falling problems and staying in supine position cause loss of motivation and decrease in quality of life for patients. In order to prevent this problem in neurological diseases, it must be evaluated and treated by working functionally as a result of this evaluation. Parkinson's patients who will participate in the study will be referred from SANKO University Sani Konukoğlu Application and Research Hospital Neurology Polyclinic. The evaluations of the patients referred from the neurology polyclinic will be carried out in SANKO University Physiotherapy and Rehabilitation Department Research Laboratory. Socio-demographic information of the included patients will be obtained. Then, the supin to stand test will be used to measure the transition time from the supine position to the standing position and mobility status, the Activity-specific balance safety scale (ABC) for fear of falling, the Berg Balance Scale for balance assessment and the timed get up and walk test, 9-hole peg test for upper extremity functionality, manual muscle testing device for muscle strength of Dorsi flexor and Plantar flexor muscle groups in the ankle, Parkinson's Disease Quality of Life Questionnaire (PHA-39) for quality of life. The evaluations to be applied will be carried out by Dr. Lecturer. Member Hakan Polat will be carried out by Hakan Polat. Apart from the supine to stand test, the other tests to be performed are tests that evaluate the parameters that an individual should have for the transition from supine to standing position. These parameters are balance, muscle strength, ability to stand up without sitting, fine motor skill ability. Supin to stand test will be re-evaluated by a different physiotherapist in SANKO University Physiotherapy and Rehabilitation Department Research Laboratory after 1 week.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is mainly caused by progressive degeneration of the nigrostriatal dopaminergic pathway and neurons in the substantia nigra pars compacta, which come together as lewy bodies or lewy neurites. PD is the most common neurodegenerative disease after Alzheimer's disease with a prevalence of 0.3% in the general population and 1-3% in the population over 65 years of age. As the disease progresses, motor and non-motor symptoms such as resting tremor, bradykinesia, rigidity, impaired reflexes, depression, anxiety, emotional changes, cognitive impairment, difficulty in swallowing, chewing and speaking, dull facial expressions, urinary problems, constipation, fatigue and sleep problems are observed with decreasing dopamine levels. In addition, people with PD usually have a flexion posture characterised by excessive thoracic kyphosis and loss of lumbar lordosis. Mobility of the neck, trunk and extremities is also lost. As the disease progresses, restrictions in bed mobility, transfers and gait can become severely disabling.

The main cause of transfer and gait problems is based on transition problems between movements. Problems such as the problem of initiating movement, freezing problem, especially when moving from one movement to another movement are very common in the later stages of Parkinson's disease. Transition problems between movements include transition from supine position to sitting position, from sitting position to standing position, from standing position to standing and walking positions. The ability to stand on the back is fundamental to people's ability to get out of bed every day. This activity is seen in neurologically affected individuals with sensoriomotor impairments, who have dynamic balance problems and muscle strength deficits, such as standing up after falls. Specific tests are needed to test this condition. We think that the supine to stand test may be valid and reliable in these individuals. If it is valid and reliable, it will be recommended to be used both in the treatment and evaluation of individuals diagnosed with Parkinson's disease. Parkinson's patients who will voluntarily participate in the study will be included. Parkinson's patients who will participate in the study will be referred from SANKO University Sani Konukoğlu Application and Research Hospital Neurology Polyclinic. The evaluations of the patients referred from the neurology polyclinic will be carried out in SANKO University Physiotherapy and Rehabilitation Department Research Laboratory. Socio-demographic information of the included patients will be obtained. Then, the supin to stand test will be used to measure the transition time from the supine position to the standing position and mobility status, the Activity-specific balance safety scale (ABC) for fear of falling, the Berg Balance Scale for balance assessment and the timed get up and walk test, 9-hole peg test for upper extremity functionality, manual muscle testing device for muscle strength of Dorsi flexor and Plantar flexor muscle groups in the ankle, Parkinson's Disease Quality of Life Questionnaire (PHA-39) for quality of life. The evaluations to be applied will be carried out by Dr. Lecturer. Member Hakan Polat will be carried out by Hakan Polat. Apart from the supine to stand test, the other tests to be performed are tests that evaluate the parameters that an individual should have for the transition from supine to standing position. These parameters are balance, muscle strength, ability to stand up without sitting, fine motor skill ability. Supin to stand test will be re-evaluated by a different physiotherapist in SANKO University Physiotherapy and Rehabilitation Department Research Laboratory after 1 week.

Demographic Information Form: This form is a form that evaluates demographic information and general information of individuals.

Supine to Stand test (SST): This test is performed to evaluate the patients' transition from supine to standing position. It measures the movement skill and how the skill is realised. For this test, we first place the patients in a supine position on a soft mat in a quiet and calm laboratory environment and ask them to stand up with the sentence 'Please stand up'. We record the time elapsed during this period. We ask the patient to repeat this test 2 times.

Activity-specific balance confidence scale (ABC) Scale: developed to measure balance confidence in indoor and outdoor activities. It is used to assess the fear of falling. It is a scale based on the respondents' assessment of how confidently they can perform 16 specified functional activities inside and outside the home on a scale from 0 (unsafe) to 100 (completely confident). The ABC scale has been shown to be a consistent and reliable method. A scale value above 80% indicates that the balance is reliable.

Timed Up and Go Test (SKYT-Timed Up and Go): Timed Up and Go (SKYT) test is a balance test frequently used to assess functional mobility in the elderly. The test measures speed during many functions such as standing, walking, turning and sitting. The test is started with the patient's feet flat on the floor and arms resting on the armrests of the chair. The test asks the person to get up from the chair (seat height 45 cm, arm height 62 cm), walk 3 metres (10ft) at a safe and usual speed, turn, walk back and sit down in the chair, and the time is recorded in seconds. A shorter time indicates better balance and mobility. In stroke patients, a test time longer than 14 seconds indicates a high risk of falling. The subjects are asked to get up as fast as possible without running, turn at the end of the road and sit down again. For the value, the timer is pressed with the start command and the time is terminated when the subject is fully seated on the chair. The elapsed time will be recorded in seconds.

Berg Balance Scale (BBS): It is one of the most basic tests that functionally evaluates balance performance in the elderly population. The scale consists of 14 functional activities frequently used in daily life (standing up while sitting, standing without support, sitting without support, sitting while standing, sitting while standing, transferring, standing with eyes closed, standing with legs together, reaching forwards while standing, picking up objects from the floor, looking backwards, turning 360 degrees, standing on a stool on the right side, standing with one foot forward and standing on one foot). The activities are scored between 0-4. If the individual cannot perform the activity, 0 points are given and 4 points are given if the individual performs the activity independently. Low scores indicate impaired balance. The highest score is 56 and 0-20 points indicate impaired balance, 21-40 points indicate the presence of an acceptable balance, 41-56 points indicate the presence of a good balance. Before starting the test, the activities will be explained to the individual one by one.9 Hole Peg Test: The 9 Hole Peg Test (9-DPT), a hand skill test, was used to evaluate fine finger skills. The test consists of a platform with 9 holes and 9 sticks. The platform was placed directly in front of the individuals and adjusted so that the rods were on the dominant hand side and the holes were on the non-dominant hand side. After the test rules were explained to the individuals, the individuals were given the opportunity to practice before the application. Individuals were asked to insert the rods on the board as fast as possible. The test results were recorded by measuring the time from the moment the individuals touched the first stick to the moment the last stick was attached to the platform with a stopwatch. Then, they were asked to remove the 9 rods one by one with the same hand and the removal time was recorded. The test will be applied for the non-dominant hand using the same method; the platform will be rotated in front of the non-dominant hand this time.

Parkinson's Quality of Life Questionnaire: Parkinson's Disease Questionnaire-39 (PDQ-39) was applied to evaluate the quality of life of the patients. PDQ-39 consists of eight sections assessing mobility, activities of daily living, mood, stigma, perception of social support, communication and body discomfort. Each section is scored separately between 0 and 100. Lower scores indicate better quality of life. For the overall assessment of quality of life, the total PDQ index can be calculated by summing the section scores. This score can also be standardised to a value between 0 and 100. Again, lower scores indicate better quality of life.

Manual muscle testing device: muscle strength (right foot dorsi flexion, left foot dorsi flexion, right foot plantar flexion, left foot plantar flexion) was measured with Commander Echo brand manual muscle testing device.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 40 years with a renewed diagnosis of Parkinson's disease
* Patients who have not changed medication in the last 2 months
* Patients who can walk with or without an assistive device

Exclusion Criteria:

* The presence of psychological or pathological conditions that can directly affect functional activity and cause metabolic changes
* Pregnant or breastfeeding women
* Alcohol and substance abusers
* Cardiovascular or metabolic disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PATIENTS WITH PARKINSON'S DISEASE ADMITTED TO THE NEUROLOGY OUTPATIENT CLINIC OF SANKO UNİVERSİTESİ SANİ KONUKOĞLU APPLICATION AND RESEARCH HOSPITAL
Sampling Method: Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Supine to Stand test (SST) | 1 Years
  This test is performed to evaluate the transition of patients from supine to standing position. It measures the movement skill and how the skill is realised. For this test, we first place the patients in a supine position on a soft mat in a quiet and calm laboratory environment and ask them to stand up with the sentence 'Please stand up'. We record the time elapsed during this period. We ask the patient to repeat this test 2 times
Activity-specific balance confidence scale (ABC) Scale | 1 Years
  developed to measure balance confidence in indoor and outdoor activities. It is used to assess the fear of falling. It is a scale based on the respondents' assessment of how confidently they can perform 16 functional activities in and out of the home, ranging from 0 (unsafe) to 100 (completely confident). The ABC scale has been shown to be a consistent and reliable method. A scale value above 80% indicates that the balance is reliable
Timed Up and Go Test (SKYT-Timed Up and Go) | 1 Years
  The Timed Up and Go (SKYT) test is a balance test frequently used to assess functional mobility in the elderly. The test measures speed during many functions such as standing, walking, turning and sitting. The test is started with the patient's feet flat on the floor and arms resting on the armrests of the chair. The test asks the person to get up from the chair (seat height 45 cm, arm height 62 cm), walk 3 metres (10ft) at a safe and usual speed, turn, walk back and sit down in the chair, and the time is recorded in seconds. A shorter time indicates better balance and mobility. In stroke patients, a test time longer than 14 seconds indicates a high risk of falling. The subjects are asked to get up as fast as possible without running, turn at the end of the road and sit down again. For the value, the timer is pressed with the start command and the time is terminated when the subject is fully seated on the chair. The elapsed time will be rec
Berg Balance Scale (BBS) | 1 Years
  is one of the most basic tests that functionally assesses balance performance in the elderly population. The scale consists of 14 functional activities frequently used in daily life (standing up while sitting, standing without support, sitting without support, sitting while standing, sitting while standing, transferring, standing with eyes closed, standing with legs together, reaching forwards while standing, picking up objects from the floor, looking backwards, turning 360 degrees, standing on a stool on the right side, standing with one foot forward and standing on one foot). Activities are scored between 0-4. If the individual cannot perform the activity, 0 points are given and 4 points are given if the individual performs the activity independently. Low scores indicate impaired balance. The highest score is 56 and 0-20 points indicate impaired balance, 21-40 points indicate the presence of an acceptable balance, 41-56 points indicate the presence of a goo
9 Hole Peg Test: | 1 years
  The 9 Hole Peg Test (9-DPT), a hand dexterity test, was used to evaluate fine finger dexterity. The test consists of a platform with 9 holes and 9 sticks. The platform was placed directly in front of the individuals and adjusted so that the rods were on the dominant hand side and the holes were on the non-dominant hand side. After the test rules were explained to the individuals, the individuals were given the opportunity to practice before the application. Individuals were asked to insert the rods on the board as fast as possible. The test results were recorded by measuring the time from the moment the individuals touched the first stick to the moment the last stick was attached to the platform with a stopwatch. Then, they were asked to remove the 9 rods one by one with the same hand and the removal time was recorded. The test will be applied for the non-dominant hand using the same method; the platform will be rotated in front of the non-dominant hand this time.
Parkinson's Quality of Life Questionnaire: | 1 Years
  Parkinson's Disease Questionnaire-39 (PDQ-39) was applied to assess the quality of life of the patients. PDQ-39 consists of eight sections assessing mobility, activities of daily living, mood, stigma, perception of social support, communication and body discomfort. Each section is scored separately between 0 and 100. Lower scores indicate better quality of life. For the overall assessment of quality of life, the total PDQ index can be calculated by summing the section scores. This score can also be standardised to a value between 0 and 100. Again, lower scores indicate better quality of life .
Manual muscle test device: | 1 Years
  muscle strength (right foot dorsi flexion, left foot dorsi flexion, right foot plantar flexion, left foot plantar flexion) will be measured with Commander Echo brand manual muscle test device. The participant will be asked to resist the resistance as much as possible and the maximum force will be recorded. After the participants are informed, 1 trial will be performed. Muscle strength measurement will be repeated 3 times and the average value will be recorded in kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- SANKO University, Gaziantep, Gazi̇azntep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
will be decided when the study is completed